CLINICAL TRIAL: NCT05314907
Title: Acceptability, Optimization and Cost-effectiveness for Self-sampling Cervical Cancer Screening.
Brief Title: Acceptability of Self-sampling for Cervical Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Collaborators: Complejo Hospitalario Universitario Insular Materno Infantil (Other); Institut Català de la Salut (Other); Institut Català d'Oncologia (Other)
Responsible Party: Principal Investigator, Raquel Ibáñez, Principal investigator, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: PI17/01179; PI17/01456 (Other Grant/Funding Number: Instituto Carlos III); PI17/01179 (Other Grant/Funding Number: Instituto Carlos III)
Record Dates: First submitted 2022-03-19; First posted 2022-04-07 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: HPV-Related Cervical Carcinoma; Self-sampling; Cervical Cancer Screening
Keywords: Self-sampling; HPV; Cervical cancer screening; Acceptability; HPV concordance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training group (Active Comparator): The Health professional shows the woman how to use the self-sampling device (Evalyn Brush) and then she collects a self-sample at the health centre as a training.
  Interventions: Device: Explanation on how to use self-sampling device and training in the screening visit.
- No prior training group (Placebo Comparator): The Health professional shows the woman how to use the self-sampling device (Evalyn Brush).
  Interventions: Other: Only explanation on how to use self-sampling device.

INTERVENTIONS:
Device: Explanation on how to use self-sampling device and training in the screening visit. — During the screening visit, woman is offered to participate in the study. If she accepts, informed consent is signed, a sociodemographic questionnaire is collected, and a cervical sample is collected for HPV detection by the health professional in the consultation.
  Then, the professional informs the woman of how to carry out the self-collection using Evalyn Brush and after the woman collects an HPV sample by self-sampling in the same medical center as a trainning.
  Finally, a new cervibrush (Evalyn brush) is given to the woman for home self-sampling, together with written and picture-based instructions on how to obtain the sample and an acceptability questionnaire. After one month from the screening visit, woman is requested to return the self-collected sample together with the questionnaire in person to the recruitment centre.
  Other Names: Evalyn Brush
  Arms: Training group
Other: Only explanation on how to use self-sampling device. — During the screening visit, woman is offered to participate in the study. If she accepts, informed consent is signed, a sociodemographic questionnaire is collected, and a cervical sample is taken for HPV detection by the health professional in the consultation.
  Then, the professional informs the woman of how to carry out the self-collection using Evalyn.
  Finally, a Evalyn brush is given to the woman for home self-sampling, together with written and picture-based instructions on how to obtain the sample and an acceptability questionnaire. After one month from the screening visit, woman is requested to return the self-collected sample together with the questionnaire in person to the recruitment centre.
  Arms: No prior training group

SUMMARY:
Main objectives:

1.1. To evaluate the use of self-sampling for HPV test in regular attendants of cervical cancer screening as a primary sample collection method.

1.2. To assess the impact on the acceptability of an educational intervention. 1.3 Confirm the concordance of HPV detection in the samples collected by the professional and in self-sampling.

Project methodology:

Randomized, parallel multicenter clinical trial in women aged 30-65 years regularly attending cervical cancer screening residents in the Autonomous Communities of Catalonia and the Canary Islands (Spain). The woman attends the routine screening visit where the health professional collects a sample from the cervical screening. She then offers her the study and if the woman accepts, she offers her the SS as a screening test. The modality of information and practice of the self-sampling is random:

1. Training group): Educational intervention with self-sampling practice: clinician-led explanation on how to proceed with self-sampling prior to collecting a self-sample at the clinic.
2. No prior trainning group): Same training without practicing self-sampling collection.

Both groups has a standard of care cervical sample collection by a clinician. Women are asked to return a self-sampling specimen one month after the baseline visit together with an acceptability questionnaire on self-sampling use.

Acceptability will be analyzed according to two definitions:

* proportion of women who returned the self-sampling device,
* proportion of women who report wanting to use self-sampling in future screens in the acceptability questionnaire.

HPV agreement between collection methods will be calculated using Cohen's Kappa coefficient. Cost-effectiveness analisis will be done on public health system by a mathematical model of the cervical cancer natural history and HPV, adjusted for data in Spain.

Self-sampling device uses in this trial is Evalyn Brush from Rovers and the HPV detection is COBAS 4800 from Roche.

DETAILED DESCRIPTION:
Women aged 30-65 years regular user of cervical cancer screening, not pregnant and with no history of cervical disease are recruited at the cervical cancer screening clinics.

Women are recruited in two Spanish distant areas, Catalonia with participant clinics in Cerdanyola del Vallés, Barberà del Vallés, Ripollet, Badia del Vallés and Sabadell, and the Canary Islands, including the clinics of Arucas, Gáldar, Prudencio Guzmán, Telde, Vecindario, Maspalomas. In both areas the cervical cancer screening was free of charge, opportunistic with cytology as primary test.

Women who agreed to participate in the study signs an informed consent and are provided with a short questionnaire including sociodemographic and screening history information.

Women are randomised, as they came to the screening visit, in two groups:

1. Training group: The trained provider shows the woman how to use the self-sampling device and asks her to collect her self-sample immediately after, at the health centre. Then, the provider gives her a new device to take a new sample at home and send it back to the health center in a month time.
2. No prior training group: The health provider shows the woman how to use self-sampling device and gives the woman a device for her to take a sample at home in a month interval and send it back to the health center.

Before the process of self-sampling, women proceed with the clinical regular screening visit. The professional collects a liquid based cervical sample. An aliquot of the sample is used for cervical cytology (screening sample) and aliquot for HPV detection (study professional sample) using the Cobas system drom Roche

The provider uses the clinical visit to explain the self-sampling process. Afterwards women in training group proceed to take her vaginal sample. In both groups a cervibrush is given for home self-sampling, together with written and picture-based instructions on how to obtain the sample and an acceptability questionnaire. After one month from the screening visit, women are requested to return the self-collected sample together with the questionnaire in person to the recruitment centre (acceptability questionnaire).

Information available for each women includes date of birth, nationality, country of birth, educational level, marital status, work, family responsibilities and data on their previous history of cervical cancer screening as if they ever did a cytology, the result of the last cytology and number of screening tests lifetime (sociodemographic questionnaire). Also, among the women who collects the self-sampling there was available information about questions on acceptability and practicalities of sampling procedures (acceptability questionnaire).

The project was approved by the ethical committees of the Bellvitge University Hospital (number PR223/17), IDIAP Jordi Gol (number P18/099) and Maternal and Child Insular University Hospital Complex (number 2018-178-1). Any information regarding the identification of patients is anonymized before analysis.

The self-sample is collected using the Rovers Medical Devices Evalyn Brush from Rovers.

Detection of HPV of all the samples from Catalonia is carried out at the Infections and Cancer laboratory of the Catalan Institute of Oncology in Barcelona, while those from the Canary Islands is processed in the Pathological Anatomy Service of the Maternal and Child Insular University Hospital Complex of Las Palmas de Gran Canaria.

All the samples are processed using Cobas HPV test Roche Cobas 4800 HPV test. Cobas HPV test is an in-vitro quantitative detection technique for high-risk HPV DNA by polymerase chain reaction (PCR) amplification and can detect a total of 14 HR-HPV subtypes and provides the results of HPV 16 and HPV 18, and the pooled results of the other 12 subtypes in the assay.

Data from both sociodemographic and acceptability questionnaires and test results (clinical and self-sampling) are collected using Research Electronic Data Capture call REDCap tools hosted at Catalan Institute of Oncology. REDCap is a secure, web-based software platform designed to support data capture for research studies, providing 1) an intuitive interface for validated data capture; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for data integration and interoperability with external sources. Personal involved in the project had access to the REDCap platform through a username and password and enter data of each woman who has been anonymized.

ELIGIBILITY:
Inclusion Criteria:

Women aged 30 to 65 years (both inclusive) with a adequate prior history of cervical cancer screening (last cytological screening test no more than four years ago).

Exclusion Criteria:

* Women under 30 years of age.
* Women over 65 years of age.
* Pregnant women.
* Women with hysterectomy.
* Women between 30 and 65 years of age who underwent the last screening test more than four years ago.
* Women between the ages of 30 and 65 who attend for follow-up of some ongoing cervical pathology.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cervical cancer screening is only for women
Enrollment: 1614 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Self-sampling acceptability for cervical cancer screening | 2 months
  Acceptability will be compared by study arm and evaluated as 1) proportion of women that return the self-sampling device, 2) proportion of women that return the self-sampling device and respond to favour future screening with self-sampling. This will be evaluated according to the sociodemographic variables of the participants and the results of the acceptability questionnaire that each woman has filled out.

SECONDARY OUTCOMES:
The cost-effectiveness of cervical Self-Sampling on public health system in Spain | This is a mathematical and cost analisis. No participants are assessed (time frame 2 years)
  A simulation model will be built based on the natural history of HPV and cervical cancer calibrated to data from Spain in reference to age-specific cervical cancer incidence and HPV prevalence. Different strategies will be evaluated that will vary according to some relevant parameters such as age and frequency of screening, self-sampling at the health center or at home. For each of the strategies, health outcomes and costs will be obtained that will allow us to calculate the reduction in lifetime cancer risk, the quality-adjusted life years (QALYs) or the cost per lifetime. Finally a cost-effectiveness analysis will be carried out between the different strategies compared to the current situation. For doing this, incremental cost-effectiveness ratios will be calculated, expressed in € per QALY gained. Finally, the impact that applying the most cost-effective interventions would have on the public health budget will be evaluated.
HPV test agreement between self-sampling and clinician-collected samples | 2 months
  A Kappa index with 95% confidence interval will be performed to observe the concordance between the HPV results from self-sampling compared to HPV results from clinical samples. A description of positivity prevalence will be also provided and the ratio of HPV positivity and the agreement (in %) between the self-sample and clinical samples will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Ibáñez Pérez, Dra., Principal Investigator — Institut Català d'Oncologia - IDIBELL; Silvia de Sanjosé Llongueras, Dra., Study Director — National Cancer Institute (NCI); Amelia Acera, Dra., Study Chair — Institut Català de la Salut; Miguel Andujar, Dr., Principal Investigator — Complejo Hospitalario Universitario Insular Materno Infantil
Locations (3):
- Spain (3):
  - Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - CAP II Cerdanyola-Ripollet - Institut Català de la Salut, Ripollet, Barcelona
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria, Canary Islands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serrano B, Ibanez R, Robles C, Peremiquel-Trillas P, de Sanjose S, Bruni L. Worldwide use of HPV self-sampling for cervical cancer screening. Prev Med. 2022 Jan;154:106900. doi: 10.1016/j.ypmed.2021.106900. Epub 2021 Nov 30. PMID 34861338
- [Derived] Ibanez R, Roura E, Acera A, Andujar M, Pavon MA, Bruni L, de Sanjose S. HPV self-sampling among cervical cancer screening users in Spain: A randomized clinical trial of on-site training to increase the acceptability. Prev Med. 2023 Aug;173:107571. doi: 10.1016/j.ypmed.2023.107571. Epub 2023 Jun 10. PMID 37308042